CLINICAL TRIAL: NCT04556227
Title: Simultaneous Recumbent Cycling and Cognitive Training on Cognition in Intensive Care Unit Survivors: a Randomized Control Trial
Brief Title: Simultaneous Recumbent Cycling and Cognitive Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri, Kansas City (Other)
Collaborators: St. Luke's Hospital, Kansas City, Missouri (Other)
Responsible Party: Principal Investigator, Rita Sue Lasiter, Associate Professor, University of Missouri, Kansas City
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 40007
Record Dates: First submitted 2020-08-24; First posted 2020-09-21 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Delirium; Impaired Cognition
Keywords: Intensive Care Unit; ICU-Survivors; Cognitive Training; Recumbent Cycling; Executive Functioning
MeSH Terms: conditions — Delirium; Cognition Disorders | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant
Masking Description: Upon leaving ICU and admission to general hospital room, study staff will go to patients' room to recruit and consent ICU survivor for study start date approximately two weeks after discharge. Randomize study participant using block randomization program. Document data on patients who decline consent and wish to be randomized to usual care or to the intervention group. This is a single masked (participant) study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Simultaneous Cycle/Cognitive Training (Experimental): After discharge from the hospital the group will engage in recumbent cycling with simultaneous cognitive training on a tablet.
  Interventions: Behavioral: Simultaneous Cycle/Cognitive Training
- Usual Care (No Intervention): After discharge from the hospital the group will complete baseline activies.

INTERVENTIONS:
Behavioral: Simultaneous Cycle/Cognitive Training — Two weeks after discharge from the hospital the intervention group will complete recumbent cycle for 1 hour, 2x/wk. for 12 weeks (24 sessions). 10-minute cycle warm-up, 40-minute simultaneous cycling and cognitive training, 10-minute cool down. Cycling based on provider prescription and progression of physical recovery. Cognitive training program from Posit Science, Brain HQ (TM) progressive level of difficulty. Total duration of 60 minutes.
  Arms: Simultaneous Cycle/Cognitive Training

SUMMARY:
Intensive care units (ICU) provide life-saving care for nearly five million people annually. Up to 80% of patients receiving care in an ICU experience at least one episode of delirium. Delirium, an acute episodic display of confused thinking and unawareness, predicts impaired cognition and accelerated cognitive decline which negatively impacts quality of life (QOL) long after hospital discharge. The average age of ICU patients is 52 years. These middle-age (MA) ICU survivors need cognitive interventions that are well planned, accessible, and effective to improve cognition and prevent accelerated decline so they can resume their previous QOL and enter older age with optimized cognitive function. Physical exercise and cognitive training independently improve cognition and emerging evidence indicates that combining these two approaches produces even greater effects on cognition. Community-based rehabilitation centers are accessible for MAICU survivors to engage in physical activity; cognitive training could easily be added. Approaches in which a patient engages in physical exercise and cognitive training concurrently is an understudied intervention for all ICU survivors, especially those who are middle-aged. Study aims are to investigate the feasibility and acceptability of a simultaneous recumbent cycling and cognitive training intervention (SRCCT) for MAICU survivors who experienced at least one delirium episode during their ICU stay. Feasibility will be determined by systematically evaluating research team training, participant recruitment, randomization, implementation, and intervention fidelity. Acceptability will be evaluated via a satisfaction, preferences, burden, and participant-suggested improvements survey. The SRCCT effect sizes will be calculated comparing multiple data point cognition scores between an SRCCT group and a usual care control group. Upon completion, investigators expect to understand the feasibility and acceptability of the SRCCT delivered in community-based rehabilitation centers, and the combined effect of SRCCT on cognition and QOL for middle-aged ICU survivors who experienced an episode of ICU delirium. The hypothesis is that study participants who engage in physical exercise and cognitive training concurrently will have a greater improvement in cognition and QOL than physical exercise training alone.

DETAILED DESCRIPTION:
Investigators will conduct a 2-year RCT, single-masked (participants), pilot feasibility and acceptability study, with repeated measures to compare SRCCT to usual care on cognition and QOL in MA, ICU survivors who experienced at least one episode of delirium in an ICU and have mild to moderate cognitive impairment. The SRCCT will include 12 weeks of simultaneous recumbent bicycling and cognitive training delivered at the same time in a rehabilitation center followed by a 6-month maintenance phase when no intervention will be delivered. Cognitive training will be administered via the POSIT Science (TM) Brain HQ computer-based program. At 12, 24, and 36 weeks post-baseline, cognition will be measured using Montreal Cognitive Assessment (MoCA) and PROMIS Cognitive Function Abilities SF8a (PRO Cog), and QOL will be assessed using PROMIS Global-10 Health Short Form (PGH-10).

Setting and Study Population: The study will take place in two large, urban health care systems in Kansas City, Missouri: St. Luke's Hospital (SLH) and Truman Medical Center (TMC). St. Luke's Hospital is located in downtown Kansas City with 600 staff physicians practicing in 60 specialty areas. This centrally located hospital has 77 ICU beds. Truman Medical Center is the safety net hospital for the Kansas City area and has 41 ICU beds. The rehabilitation centers employ healthcare staff who work with outpatients who are deconditioned and recovering from hospitalization. Data provided by SLH and TMC indicate an adequate pool for study recruitment. In 2018, 87 MA patients were admitted to TMC ICUs; 1366 were admitted to SLH ICUs. Combined ICU admissions age 45-64 were 1453 and 12% (174) experienced delirium (using CAM-ICU). Given 79% (138) of patients who have ICU delirium experience cognitive impairment and recruitment rate of 75%, there are 103 ICU survivors possible and therefore the recruitment goal of 50 participants for this study is achievable. Fifty patients meeting inclusion criteria will be recruited and enrolled.The final patient sample will comprise 50 MA ICU survivors who have had at least one episode of delirium in the ICU and have mild to moderate cognitive impairment (using MoCA). Registered Nurses (RN) from SLH and TM CICUs will identify and HIPAA-consent patients who meet study inclusion and exclusion criteria. Once consented, the RN will notify the study Research Assistant (RA). After discharge from the ICU to a hospital room, the RA will meet with the patient to explain the study and obtain consent. Once consented, the RA will contact the PI's who will determine random assignment to either treatment (SRCCT) or usual care. Block randomization will be created using a computer-generated list of random numbers blocked into balanced groups of four. Before recruitment begins, the RAs will practice the consent process in simulated situations with PIs. Rapport will be maintained by pairing RAs and participants for the duration of the intervention thereby enhancing retention. Investigators anticipate low attrition but recognize participants may withdraw 1) on the advice of their healthcare provider or for other health reasons, 2) due to changes in life circumstances, or 3) loss of interest in the study. In such cases, the RAs will document the event and notify the PIs who will track all withdrawals. Patients who are randomized to the SRCCT intervention treatment group will be screened and consented after transition from ICU into their hospital room. The SRCCT will begin approximately two weeks after discharge to home. The intervention was developed by Dr. Lasiter (Co-PI and Critical Care nurse), Dr. Chrisman (Co-PI and physical activity interventionist), and Dr. Russell (Co-I and feasibility/acceptability/RCT expert) and will be administered by Drs. Lasiter and Chrisman, and two trained RAs. A rehabilitation center RN will monitor the participant's condition while engaged in the SRCCT or usual care. Dr. Lasiter and Dr. Chrisman will oversee the intervention protocol. Research assistants who are baccalaureate and master's-prepared RNs experienced in RCT studies will undergo training by Drs. Lasiter, Chrisman, and Russell, including the following components: 1) project rationale and overview; 2) detailed information on the SRCCT intervention and usual care; 3) scripts for use when consenting and collecting data; 4) how to use Research Electronic Data Capture (REDCap) database (redcap.umkc.edu); 5) detailed training on administering study instruments (MoCA requires training before permission is granted to use the instrument), and 6) using a tablet. Simulation and role-play will be used until the RAs are consistently applying the protocol as judged by investigators. To ensure the highest level of RA protocol knowledge and skills, the training sessions will also include role-playing of disruptive situations for the intervention. To monitor RA intervention fidelity, a fidelity protocol checklist will be used during all participant encounters to document key elements of the protocol, including number of intervention sessions, session duration, length of time between sessions, and intervention steps. Each element will be rated as completed, partially completed, not completed, or N/A. Field notes will be kept for every encounter. Participants randomized into the usual care arm will receive scheduled follow-up office appointments with their provider post-discharge at which time a member of the study team will administer the scheduled study measures at specific time points. The usual care group will not receive SRCCT.

Data analyses: Drs. Lasiter, Chrisman and Staggs (biostatistician) will conduct analyses. Feasibility will be tracked using checklists for 1) educating nursing staff about inclusion criteria and HIPAA consent, 2) educating RAs about interpersonal communication, recruitment, consent, intervention procedures and fidelity and, 3) guiding the intervention to insure fidelity between sites and study staff/investigators. Acceptability will be evaluated by assessing four domains: participant satisfaction, participant preferences, participant burden, and suggestions for improvement. Limitations: One limitation is that the study will not include exercise-only or cognitive-only training groups. Literature supports that each is effective independently and, rather than isolate their effects, investigators will examine combined effects which has the potential to be synergistic in efficacy. Potential difficulty may be recruitment; if recruitment difficulty occurs, investigators will consult with the study team and study site contacts to potentially widen the scope of recruiting participants, add a third study site, or hire an RA who closely matches the ages of the study sample. Another potential difficulty is low retention, and/or patient mortality. To minimize attrition, an honoraria will be provided for each data collection time point. Although mortality in MA ICU survivors is higher than in the general MA population, investigators do not expect mortality to have a major effect on retention in this 36-week study.

Data Analyses Plan: Descriptive statistics (e.g., standardized mean difference) will be used to compare the intervention and control groups on selected patient characteristics and adjust for meaningful imbalances on any variables by including them as covariates in statistical modeling. In the focal analysis investigators will assess the effect of the SRCCT intervention on each of the three Aim 1 outcome measures at T3 by fitting three ANCOVA models with the T3 measurement as the dependent variable, the baseline measurement (T2) as a covariate, and group (intervention vs. control) as an explanatory variable. In secondary analyses the intervention effect at T4 and T5 will be assessed analogously. If the usual linear modeling assumption of Normal residuals is not met, investigators will either transform the dependent variable, fit an appropriate generalized linear model, or obtain confidence limits and p-values by non-parametric bootstrapping. Power and precision of estimation for the ANCOVA model described above were assessed using a simulation study. For each of 1,000 simulated data sets, investigators randomly generated Normal T2 scores and then used these to generate Normal T3 scores, assuming a strong intervention effect of 0.5 SDs and a correlation of 0.7 between T2 and T3 scores within each arm (implying roughly 50% of variability in T3 scores can be explained by T2 scores). In keeping with the exploratory nature of this aim, power was estimated to detect a non-zero intervention effect with a one-sided test at α = 0.10. The average length of the 90% confidence interval for the intervention effect across the simulated data sets was computed. Estimated power was 86%, and confidence intervals averaged 0.68 SDs in length (equivalent to an average margin of error of 0.34 SDs). Actual power will depend on the true intervention effect size and true correlation between T2 and T3 scores, both of which are unknown; however, in this preliminary effort to demonstrate efficacy the focus will be on estimating the intervention effect size, not making a yes/no decision in a null hypothesis test based on an arbitrary α cutoff. Analyses will be run using an intent-to-treat approach, with missing data addressed either by multiple imputation or nonresponse weighting.

ELIGIBILITY:
Inclusion Criteria:

* Age 45-64 years
* Admitted to medical or surgical ICUs (SLH & TMC) for >24 hours
* English-speaking
* Discharged home
* Able to provide consent
* Access to a telephone
* One or more delirium episode in ICU (positive CAM-ICU).

Exclusion Criteria:

* Cancer diagnosis with short life expectancy determined by the Primary Care Provider (unable to complete the study within time frame)
* Chemotherapy (drug-induced impaired cognition)
* Diagnosed vascular dementia or other neurodegenerative diseases (e.g. Alzheimer or Parkinson disease)
* Documented alcohol consumption ≥5 drinks/day (withdrawal delirium tremens)
* Corrected vision<20/80 Snellen chart (unable to do cognitive exercises on the tablet)
* Examiner rated low hearing or communicative ability that would interfere with intervention and assessments
* Positive CAM-ICU (delirium) at hospital discharge
* Unable to participate in rehabilitation (abnormal 6 min walk test)
* Any physical condition preventing recumbent cycling
* Recent documented history of drug abuse.

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-03 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Simultaneous Recumbent Cycling and Cognitive Training Survey | At study completion, approximately 36 weeks.
  Feasibility of participant recruitment, randomization, intervention, intervention fidelity, and data collection. Less problems to overcome with recruitment, randomization, administering intervention, and data collection the more feasible the study.
Acceptability of Simultaneous Recumbent Cycling and Cognitive Training Survey | Approximately 24 weeks.
  Acceptability Survey: Determine satisfaction and burden including text suggestions for study improvement. Likert type scale 1-4; higher score means more acceptable.

SECONDARY OUTCOMES:
Change in Cognition using Montreal Cognitive Assessment Test | Screening for inclusion, 2 weeks,12 weeks, 24 weeks, and at study completion, approximately 36 weeks.
  Cognitive status assessed at multiple data collection points using the Montreal Cognitive Assessment Test. The following composite scores may be used to grade severity: 18-25 = mild cognitive impairment, 10-17= moderate cognitive impairment and less than 10= severe cognitive impairment.
Change in perceived cognition using Patient-Reported Outcomes Measurement Information System, Applied Cognition Short Form-8. | Baseline,12 weeks, 24 weeks, and at study completion, approximately 36 weeks.
  Participants' perception of daily cognition using the Patient-Reported Outcomes Measurement Information System (PROMIS), Applied Cognition Short Form-8 item and composite scores; higher score means better outcome.
Quality of life using Patient-Reported Outcomes Measurement Information System Global-10 Short Form | Baseline,12 weeks, and at study completion, approximately 36 weeks.
  Patient-Reported Outcomes Measurement Information System (PROMIS) Global-10 Short Form used to measure physical, mental, and social health quality of life. Item and composite score; higher score means better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Rita S Lasiter, PhD, Principal Investigator — University of Missouri, Kansas City; Matthew S Chrisman, PhD, Principal Investigator — University of Missouri, Kansas City
Locations (1):
- St. Luke's Hospital of Kansas City, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Utilization of Intensive Care Services, 2011 #185. https://hcup-us.ahrq.gov/reports/statbriefs/sb185-Hospital-Intensive-Care-Units-2011.jsp. Accessed September 2, 2019.
- [Background] Needham DM, Davidson J, Cohen H, Hopkins RO, Weinert C, Wunsch H, Zawistowski C, Bemis-Dougherty A, Berney SC, Bienvenu OJ, Brady SL, Brodsky MB, Denehy L, Elliott D, Flatley C, Harabin AL, Jones C, Louis D, Meltzer W, Muldoon SR, Palmer JB, Perme C, Robinson M, Schmidt DM, Scruth E, Spill GR, Storey CP, Render M, Votto J, Harvey MA. Improving long-term outcomes after discharge from intensive care unit: report from a stakeholders' conference. Crit Care Med. 2012 Feb;40(2):502-9. doi: 10.1097/CCM.0b013e318232da75. PMID 21946660
- [Background] Ely EW, Inouye SK, Bernard GR, Gordon S, Francis J, May L, Truman B, Speroff T, Gautam S, Margolin R, Hart RP, Dittus R. Delirium in mechanically ventilated patients: validity and reliability of the confusion assessment method for the intensive care unit (CAM-ICU). JAMA. 2001 Dec 5;286(21):2703-10. doi: 10.1001/jama.286.21.2703. PMID 11730446
- [Background] Khan BA, Lasiter S, Boustani MA. CE: critical care recovery center: an innovative collaborative care model for ICU survivors. Am J Nurs. 2015 Mar;115(3):24-31; quiz 34, 46. doi: 10.1097/01.NAJ.0000461807.42226.3e. PMID 25674682
- [Background] Desai SV, Law TJ, Needham DM. Long-term complications of critical care. Crit Care Med. 2011 Feb;39(2):371-9. doi: 10.1097/CCM.0b013e3181fd66e5. PMID 20959786
- [Background] Rothenhausler HB, Ehrentraut S, Stoll C, Schelling G, Kapfhammer HP. The relationship between cognitive performance and employment and health status in long-term survivors of the acute respiratory distress syndrome: results of an exploratory study. Gen Hosp Psychiatry. 2001 Mar-Apr;23(2):90-6. doi: 10.1016/s0163-8343(01)00123-2. PMID 11313077
- [Background] Pandharipande PP, Girard TD, Jackson JC, Morandi A, Thompson JL, Pun BT, Brummel NE, Hughes CG, Vasilevskis EE, Shintani AK, Moons KG, Geevarghese SK, Canonico A, Hopkins RO, Bernard GR, Dittus RS, Ely EW; BRAIN-ICU Study Investigators. Long-term cognitive impairment after critical illness. N Engl J Med. 2013 Oct 3;369(14):1306-16. doi: 10.1056/NEJMoa1301372. PMID 24088092
- [Background] Griffiths J, Hatch RA, Bishop J, Morgan K, Jenkinson C, Cuthbertson BH, Brett SJ. An exploration of social and economic outcome and associated health-related quality of life after critical illness in general intensive care unit survivors: a 12-month follow-up study. Crit Care. 2013 May 28;17(3):R100. doi: 10.1186/cc12745. PMID 23714692
- [Background] Kamdar BB, Huang M, Dinglas VD, Colantuoni E, von Wachter TM, Hopkins RO, Needham DM; National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome Network. Joblessness and Lost Earnings after Acute Respiratory Distress Syndrome in a 1-Year National Multicenter Study. Am J Respir Crit Care Med. 2017 Oct 15;196(8):1012-1020. doi: 10.1164/rccm.201611-2327OC. PMID 28448162
- [Background] Norman BC, Jackson JC, Graves JA, Girard TD, Pandharipande PP, Brummel NE, Wang L, Thompson JL, Chandrasekhar R, Ely EW. Employment Outcomes After Critical Illness: An Analysis of the Bringing to Light the Risk Factors and Incidence of Neuropsychological Dysfunction in ICU Survivors Cohort. Crit Care Med. 2016 Nov;44(11):2003-2009. doi: 10.1097/CCM.0000000000001849. PMID 27171492
- [Background] Tropea J, LoGiudice D, Liew D, Gorelik A, Brand C. Poorer outcomes and greater healthcare costs for hospitalised older people with dementia and delirium: a retrospective cohort study. Int J Geriatr Psychiatry. 2017 May;32(5):539-547. doi: 10.1002/gps.4491. Epub 2016 Apr 25. PMID 27114271
- [Background] Zhu X, Yin S, Lang M, He R, Li J. The more the better? A meta-analysis on effects of combined cognitive and physical intervention on cognition in healthy older adults. Ageing Res Rev. 2016 Nov;31:67-79. doi: 10.1016/j.arr.2016.07.003. Epub 2016 Jul 14. PMID 27423932
- [Background] Bruderer-Hofstetter M, Rausch-Osthoff AK, Meichtry A, Munzer T, Niedermann K. Effective multicomponent interventions in comparison to active control and no interventions on physical capacity, cognitive function and instrumental activities of daily living in elderly people with and without mild impaired cognition - A systematic review and network meta-analysis. Ageing Res Rev. 2018 Aug;45:1-14. doi: 10.1016/j.arr.2018.04.002. Epub 2018 Apr 18. PMID 29679658
- [Background] Lasiter S, Snodgrass B, Thompson M, Chrisman M. Physical activity and cognitive training as interventions to enhance cognitive functioning: A systematic review. unpublished manuscript.
- [Background] Northey JM, Cherbuin N, Pumpa KL, Smee DJ, Rattray B. Exercise interventions for cognitive function in adults older than 50: a systematic review with meta-analysis. Br J Sports Med. 2018 Feb;52(3):154-160. doi: 10.1136/bjsports-2016-096587. Epub 2017 Apr 24. PMID 28438770
- [Background] Gross AL, Parisi JM, Spira AP, Kueider AM, Ko JY, Saczynski JS, Samus QM, Rebok GW. Memory training interventions for older adults: a meta-analysis. Aging Ment Health. 2012;16(6):722-34. doi: 10.1080/13607863.2012.667783. PMID 22423647
- [Background] Jackson JC, Ely EW, Morey MC, Anderson VM, Denne LB, Clune J, Siebert CS, Archer KR, Torres R, Janz D, Schiro E, Jones J, Shintani AK, Levine B, Pun BT, Thompson J, Brummel NE, Hoenig H. Cognitive and physical rehabilitation of intensive care unit survivors: results of the RETURN randomized controlled pilot investigation. Crit Care Med. 2012 Apr;40(4):1088-97. doi: 10.1097/CCM.0b013e3182373115. PMID 22080631
- [Background] Ohman H, Savikko N, Strandberg TE, Pitkala KH. Effect of physical exercise on cognitive performance in older adults with mild cognitive impairment or dementia: a systematic review. Dement Geriatr Cogn Disord. 2014;38(5-6):347-65. doi: 10.1159/000365388. Epub 2014 Aug 21. PMID 25171577
- [Background] Yu F, Kolanowski A. Facilitating aerobic exercise training in older adults with Alzheimer's disease. Geriatr Nurs. 2009 Jul-Aug;30(4):250-9. doi: 10.1016/j.gerinurse.2008.11.001. Epub 2009 Mar 9. PMID 19665667
- [Background] Brummel NE, Girard TD, Ely EW, Pandharipande PP, Morandi A, Hughes CG, Graves AJ, Shintani A, Murphy E, Work B, Pun BT, Boehm L, Gill TM, Dittus RS, Jackson JC. Feasibility and safety of early combined cognitive and physical therapy for critically ill medical and surgical patients: the Activity and Cognitive Therapy in ICU (ACT-ICU) trial. Intensive Care Med. 2014 Mar;40(3):370-9. doi: 10.1007/s00134-013-3136-0. Epub 2013 Nov 21. PMID 24257969
- [Background] Leavell HR, Clark EG. Textbook of Preventive Medicine. New York: McGraw-Hill; 1953
- [Background] Leavell HR, Clark EG. Preventive Medicine for the Doctor in His Community, An Epidemiological Approach. 2nd ed. New York: McGraw-Hill; 1958.
- [Background] Berney S, Haines K, Skinner EH, Denehy L. Safety and feasibility of an exercise prescription approach to rehabilitation across the continuum of care for survivors of critical illness. Phys Ther. 2012 Dec;92(12):1524-35. doi: 10.2522/ptj.20110406. Epub 2012 Aug 9. PMID 22879441
- [Background] Shields GE, Wells A, Doherty P, Heagerty A, Buck D, Davies LM. Cost-effectiveness of cardiac rehabilitation: a systematic review. Heart. 2018 Sep;104(17):1403-1410. doi: 10.1136/heartjnl-2017-312809. Epub 2018 Apr 13. PMID 29654096
- [Background] Denehy L, Skinner EH, Edbrooke L, Haines K, Warrillow S, Hawthorne G, Gough K, Hoorn SV, Morris ME, Berney S. Exercise rehabilitation for patients with critical illness: a randomized controlled trial with 12 months of follow-up. Crit Care. 2013 Jul 24;17(4):R156. doi: 10.1186/cc12835. PMID 23883525
- [Background] Lasiter S, Oles SK, Mundell J, London S, Khan B. Critical Care Follow-up Clinics: A Scoping Review of Interventions and Outcomes. Clin Nurse Spec. 2016 Jul-Aug;30(4):227-37. doi: 10.1097/NUR.0000000000000219. PMID 27309787
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] PROMIS: Clinical Outcomes Assessment. https://commonfund.nih.gov/promis/index. Accessed September 7, 2019.
- [Background] Ouimet S, Kavanagh BP, Gottfried SB, Skrobik Y. Incidence, risk factors and consequences of ICU delirium. Intensive Care Med. 2007 Jan;33(1):66-73. doi: 10.1007/s00134-006-0399-8. Epub 2006 Nov 11. PMID 17102966
- [Background] Milbrandt EB, Deppen S, Harrison PL, Shintani AK, Speroff T, Stiles RA, Truman B, Bernard GR, Dittus RS, Ely EW. Costs associated with delirium in mechanically ventilated patients. Crit Care Med. 2004 Apr;32(4):955-62. doi: 10.1097/01.ccm.0000119429.16055.92. PMID 15071384
- [Background] Zhao J, Yao L, Wang C, Sun Y, Sun Z. The effects of cognitive intervention on cognitive impairments after intensive care unit admission. Neuropsychol Rehabil. 2017 Apr;27(3):301-317. doi: 10.1080/09602011.2015.1078246. Epub 2015 Aug 27. PMID 26313129
- [Background] Zheng G, Xia R, Zhou W, Tao J, Chen L. Aerobic exercise ameliorates cognitive function in older adults with mild cognitive impairment: a systematic review and meta-analysis of randomised controlled trials. Br J Sports Med. 2016 Dec;50(23):1443-1450. doi: 10.1136/bjsports-2015-095699. Epub 2016 Apr 19. PMID 27095745
- [Background] Karssemeijer EGA, Aaronson JA, Bossers WJ, Smits T, Olde Rikkert MGM, Kessels RPC. Positive effects of combined cognitive and physical exercise training on cognitive function in older adults with mild cognitive impairment or dementia: A meta-analysis. Ageing Res Rev. 2017 Nov;40:75-83. doi: 10.1016/j.arr.2017.09.003. Epub 2017 Sep 12. PMID 28912076
- [Background] Vaportzis E, Niechcial MA, Gow AJ. A systematic literature review and meta-analysis of real-world interventions for cognitive ageing in healthy older adults. Ageing Res Rev. 2019 Mar;50:110-130. doi: 10.1016/j.arr.2019.01.006. Epub 2019 Jan 29. PMID 30707947
- [Background] Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, McLeod L, Delacqua G, Delacqua F, Kirby J, Duda SN; REDCap Consortium. The REDCap consortium: Building an international community of software platform partners. J Biomed Inform. 2019 Jul;95:103208. doi: 10.1016/j.jbi.2019.103208. Epub 2019 May 9. PMID 31078660
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Hamilton DM, Haennel RG. Validity and reliability of the 6-minute walk test in a cardiac rehabilitation population. J Cardiopulm Rehabil. 2000 May-Jun;20(3):156-64. doi: 10.1097/00008483-200005000-00003. PMID 10860197
- [Background] Saffer BY, Lanting SC, Koehle MS, Klonsky ED, Iverson GL. Assessing cognitive impairment using PROMIS((R)) applied cognition-abilities scales in a medical outpatient sample. Psychiatry Res. 2015 Mar 30;226(1):169-72. doi: 10.1016/j.psychres.2014.12.043. Epub 2015 Jan 8. PMID 25639374
- [Background] Howland M, Tatsuoka C, Smyth KA, Sajatovic M. Evaluating PROMIS((R)) applied cognition items in a sample of older adults at risk for cognitive decline. Psychiatry Res. 2017 Jan;247:39-42. doi: 10.1016/j.psychres.2016.10.072. Epub 2016 Nov 1. PMID 27863317
- [Background] Hays RD, Bjorner JB, Revicki DA, Spritzer KL, Cella D. Development of physical and mental health summary scores from the patient-reported outcomes measurement information system (PROMIS) global items. Qual Life Res. 2009 Sep;18(7):873-80. doi: 10.1007/s11136-009-9496-9. Epub 2009 Jun 19. PMID 19543809